CLINICAL TRIAL: NCT04508023
Title: A Multicenter, Randomized, Placebo-Controlled, Pragmatic Phase 3 Study Investigating the Efficacy and Safety of Rivaroxaban to Reduce the Risk of Major Venous and Arterial Thrombotic Events, Hospitalization and Death in Medically Ill Outpatients With Acute, Symptomatic COVID-19 Infection
Brief Title: A Study of Rivaroxaban to Reduce the Risk of Major Venous and Arterial Thrombotic Events, Hospitalization and Death in Medically Ill Outpatients With Acute, Symptomatic Coronavirus Disease 2019 (COVID-19) Infection
Acronym: PREVENT-HD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prematurely due to enrollment challenges.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108849; 39039039DVT3004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Participants will receive rivaroxaban 10 milligram (mg) tablet orally once daily for 35 Days along with standard of care treatment (SOC).
  Interventions: Drug: Rivaroxaban; Other: Standard of Care (SOC)
- Placebo (Placebo Comparator): Participants will receive matching placebo tablet orally once daily for 35 Days along with SOC.
  Interventions: Other: Placebo; Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Rivaroxaban — Participants will receive rivaroxaban 10 mg tablet orally once daily.
  Other Names: JNJ-39039039; BAY 59-7939
  Arms: Rivaroxaban
Other: Placebo — Participants will receive matching placebo tablet orally once daily.
  Arms: Placebo
Other: Standard of Care (SOC) — SOC treatment will be determined by the investigator based on local practice and consists of supportive care.

SUMMARY:
The purpose of this study is to evaluate whether rivaroxaban reduces the risk of a composite endpoint of major venous and arterial thrombotic events, all-cause hospitalization, and all-cause mortality compared with placebo in outpatients with acute, symptomatic Coronavirus Disease 2019 (COVID-19) Infection.

ELIGIBILITY:
Inclusion Criteria:

* Coronavirus Disease 2019 (COVID-19) positive diagnosis by locally obtained viral diagnostic test (example, polymerase chain reaction [PCR]). This may be nasal swab or saliva test or other available technology to demonstrate current infection
* Confirm that participant is known to health system, with at least 1 contact in electronic medical records (EMR) prior to screening
* Symptoms attributable to COVID-19 (example, fever, cough, loss of taste or smell, muscle aches, shortness of breath, fatigue)
* Initial treatment plan does not include hospitalization
* Presence of at least 1 additional risk factor: a) age more than or equal to (>=) 60 years; b) prior history of VTE; c) history of thrombophilia; d) history of coronary artery disease (CAD); e) history of peripheral artery disease (PAD); f) history of cerebrovascular disease or ischemic stroke; g) history of cancer (other than basal cell carcinoma) h) history of diabetes requiring medication; i) history of heart failure; j) body mass index (BMI) greater than or equal to (>=) 35 kilogram per meter square (kg/m^2); k) D-dimer greater than (>) upper limit of normal for local laboratory (within 2 weeks of the date of the COVID-19 test and prior to randomization)

Exclusion Criteria:

* Increased risk of bleeding such as a) significant bleeding in the last 3 months; b) active gastroduodenal ulcer in the last 3 months; c) history of bronchiectasis or pulmonary cavitation; d) need for dual antiplatelet therapy or anticoagulation; e) prior intracranial hemorrhage, f) known severe thrombocytopenia g) active cancer and undergoing treatment
* Any illness or condition that in the opinion of the investigator would significantly increase the risk of bleeding (example recent trauma, recent surgery, severe uncontrolled hypertension, gastrointestinal cancer, renal failure requiring dialysis, severe liver disease, known bleeding diathesis)
* Known allergies, hypersensitivity, or intolerance to rivaroxaban or its excipients
* Positive COVID-19 antibody or serology test after 2-week period of acute, symptomatic COVID-19 infection
* Known diagnosis of triple positive (positive for lupus anticoagulant, anticardiolipin, and anti-beta 2-glycoprotein I antibodies) antiphospholipid syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1284 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (17):
  - University of Arizona, Tucson, Arizona
  - Southern California Permanente Medical Group, Los Angeles, California
  - Kaiser Permanente Northern California, Oakland, California
  - University of Colorado Denver, Aurora, Colorado
  - Florida Hospital Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northshore Universite Healthsystem, Evanston, Illinois
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Lenox Hill Hospital -Northwell Health, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Health Physicians Group, Fort Worth, Texas
  - Franciscan Research Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Result] Piazza G, Spyropoulos AC, Hsia J, Goldin M, Towner WJ, Go AS, Bull TM, Weng S, Lipardi C, Barnathan ES, Bonaca MP; PREVENT-HD Investigators. Rivaroxaban for Prevention of Thrombotic Events, Hospitalization, and Death in Outpatients With COVID-19: A Randomized Clinical Trial. Circulation. 2023 Jun 20;147(25):1891-1901. doi: 10.1161/CIRCULATIONAHA.123.063901. Epub 2023 May 8. PMID 37154020
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were not treated with study drug were still followed-up as per the planned visits.
Groups:
- Rivaroxaban 10 Milligrams (mg): Eligible participants with symptomatic coronavirus disease 2019 (COVID-19) who were at risk of venous and arterial thrombotic complications, received rivaroxaban 10 mg, orally, once daily throughout the 35 days of double-blind treatment period along with ongoing standard of care medications for COVID-19 at the discretion of the treating physician.
- Placebo: Eligible participants with symptomatic COVID-19 who were at risk of venous and arterial thrombotic complications, received placebo matching to rivaroxaban, orally, once daily throughout the 35 days of double-blind treatment period along with ongoing standard of care medications for COVID-19 at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
Started | 641 | 643
Treated (Safety Analysis Set) | 599 | 598
Completed (This also included participants who were not treated with study drug, but were still followed-up as per the planned visits.) | 640 | 641
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo | Total
Number analyzed (Participants) | 641 | 643 | 1284
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.07) | 55.7 (13.3) | 56 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 399 | 384 | 783
  Male | 242 | 259 | 501
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 97 | 192
  Not Hispanic or Latino | 520 | 508 | 1028
  Unknown or Not Reported | 26 | 38 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 25 | 16 | 41
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 61 | 65 | 126
  White | 465 | 464 | 929
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 85 | 90 | 175
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 641 | 643 | 1284

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Time to First Occurrence of Primary Efficacy Composite Endpoint
Description: Number of participants with time to first occurrence of primary efficacy composite endpoint were reported. Time to first occurrence of primary efficacy composite endpoint is defined as time from randomization to first occurrence of any component of the primary endpoint. The components were: symptomatic venous thromboembolism (VTE), myocardial infarction (MI), ischemic stroke, acute limb ischemia, non-central nervous system (non-CNS) systemic embolization, all-cause hospitalization, and all-cause mortality.
Time Frame: Up to Day 35
Population: Intent-To-Treat (ITT) analysis set included all randomized participants who provided informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 641 | 643
Participants | 22 | 19
Statistical Analysis 1: Comparison: Rivaroxaban 10 Milligrams (mg) vs Placebo; Test type: Superiority; p = 0.626, Log Rank; Log rank test stratified by the time from COVID-19 positive test to randomization; Cox Proportional Hazard = 1.16, 95% CI 2-sided [0.63 to 2.15]

2. Primary Outcome: Number of Participants With Time to First Occurrence of The Principle Safety Outcome (Fatal Bleeding and Critical Site Bleeding) Based on a Modification of the International Society on Thrombosis and Haemostasis (ISTH) Criteria
Description: Number of participants with time to first occurrence of the principle safety outcome (fatal bleeding and critical site bleeding) based on a Modification of the ISTH criteria were reported. Fatal bleeding is defined as any bleeding event that leads to fatal outcome. Critical site bleeding defined as any bleeding event that occurred at critical site such as intracranial, intra-spinal, intraocular, pericardial, intra-articular, intra-muscular with compartment syndrome, retroperitoneal.
Time Frame: Up to Day 35
Population: The safety analysis set included participants in ITT who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 599 | 598
Participants
  Fatal Bleeding | 0 | 0
  Critical Site Bleeding | 0 | 0

3. Secondary Outcome: Number of Participants With Time to the First Occurrence of Secondary Efficacy Outcomes
Description: Number of participants with time to the first occurrence of secondary efficacy outcomes which included thrombotic events (symptomatic VTE, myocardial infarction, ischemic stroke, acute limb ischemia, non-CNS systemic embolization), emergency room (ER) visit, all-cause mortality, all-cause hospitalization, any thrombotic outcome and all-cause mortality, and any thrombotic outcome and all-cause hospitalization, were reported.
Time Frame: From Day 1 up to Day 35
Population: ITT analysis set included all randomized participants who provided informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 641 | 643
Participants
  Symptomatic VTE | 0 | 3
  Myocardial Infraction | 0 | 0
  Ischemic stroke | 0 | 2
  Acute limb ischemia | 0 | 0
  Non-CNS systemic embolization | 0 | 0
  ER Visit | 26 | 34
  All-cause hospitalization | 21 | 17
  All-cause Mortality | 2 | 2
  Any Thrombotic Outcome and All-cause Mortality | 2 | 7
  Any Thrombotic Outcome and All-cause Hospitalization | 21 | 17

4. Secondary Outcome: Number of Participants With Time to First Occurrence of Major Bleeding Based on a Modification of the ISTH Criteria
Description: Number of participants with time to first occurrence of the major bleeding based on a modification of the ISTH criteria were reported. Major bleeding is defined as clinically overt bleeding that is associated with a reduction in hemoglobin of 2 grams per deciliter (g/dL) or more, or a transfusion of 2 or more units of packed red blood cells or whole blood, or occurrence at a critical site defined as intracranial, intra-spinal, intraocular, pericardial, intra-articular, intra-muscular with compartment syndrome, retroperitoneal, or fatal outcome.
Time Frame: Up to Day 35
Population: The safety analysis set included participants in ITT who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 599 | 598
Participants | 1 | 0

5. Secondary Outcome: Number of Participants Who Were Hospitalized or Dead on Day 35
Description: Number of participants who were hospitalized or dead on Day 35 were reported.
Time Frame: At Day 35 (+/- 6 days)
Population: ITT analysis set included all randomized participants who provided informed consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
Number analyzed (Participants) | 641 | 643
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: Adverse Event collection started from screening up to Day 49 post-treatment follow-up
Description: All-cause mortality was analyzed based on intent-to-treat (ITT) set defined as all randomized participants who provided informed consent. Serious adverse events and other adverse events were analyzed based on the safety analysis set defined as all participants who received at least 1 dose of study intervention.
Arm/Group | Rivaroxaban 10 Milligrams (mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/641 | 2/643
Serious Adverse Events (participants affected / at risk) | 1/599 | 0/598
Other Adverse Events (participants affected / at risk) | 57/599 | 50/598
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 10 Milligrams (mg) (N=599) | Placebo (N=598)
Drug Hypersensitivity (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban 10 Milligrams (mg) (N=599) | Placebo (N=598)
Angina Pectoris (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 2
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Eye Pruritus (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Dry Mouth (Gastrointestinal disorders) | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Feeling Hot (General disorders) | 1 | 0
Injection Site Bruising (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Peripheral Swelling (General disorders) | 1 | 0
Vaccination Site Bruising (General disorders) | 0 | 1
Allergy to Animal (Immune system disorders) | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 3 | 2
Ear Infection (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pharyngitis Streptococcal (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Liver Function Test Increased (Investigations) | 0 | 1
Oxygen Saturation Decreased (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2
Dizziness Exertional (Nervous system disorders) | 1 | 0
Dizziness Postural (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Restless Legs Syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Irritability (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 0 | 1
Polycystic Ovaries (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Blood Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Peripheral Coldness (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to enrollment challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT04508023/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04508023/SAP_003.pdf